CLINICAL TRIAL: NCT04267276
Title: Investigation of Metabolism and Pharmacokinetics of BI 1265162 (C-14) After Intravenous Administration (Part 1) and Investigation of Metabolism and Pharmacokinetics of BI 1265162 (C-14) After Oral Administration (Part 2) in Healthy Male Subjects Following a Non-randomized, Open-label, Single-dose, Single Arm Per Trial Part Mass Balance Design
Brief Title: A Study in Healthy Men to Test How BI 1265162 is Taken up and Processed by the Body
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to the COVID-19 pandemic, the recruitment of new subjects was temporarily halted in March 2020. The study was permanently discontinued in December 2020.
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1399-0013; 2019-003389-42 (EudraCT Number)
Record Dates: First submitted 2020-02-11; First posted 2020-02-12 (Actual); Results first posted 2022-02-23 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: BI 1265162 - intravenous (Experimental)
  Interventions: Drug: Part 1: BI 1265162 - intravenous
- Part 2: BI 1265162 - oral (Experimental)
  Interventions: Drug: Part 2: BI 1265162 - oral

INTERVENTIONS:
Drug: Part 1: BI 1265162 - intravenous — Intravenous solution
  Arms: Part 1: BI 1265162 - intravenous
Drug: Part 2: BI 1265162 - oral — Oral solution
  Arms: Part 2: BI 1265162 - oral

SUMMARY:
To investigate rates and routes of excretion, mass balance, pharmacokinetics of parent drug, any known metabolites, and total radioactivity, metabolite profiling, metabolite identification, if suitable assays are available, safety and tolerability in healthy male subjects.

ELIGIBILITY:
Inclusion criteria

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocrdiogram (ECG), and clinical laboratory tests
* Age of 18 to 65 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the trial, in accordance with Good Clinical Practice (GCP) and local legislation
* Subjects who are sexually active must use, with their partner, highly effective contraception from the time of administration of trial medication until 3 months after administration of trial medication. Adequate methods are:

  * Condoms plus use of hormonal contraception by the female partner that started at least 2 months prior to administration of trial medication (e.g., implants, injectables, combined oral or vaginal contraceptives, intrauterine device), or
  * Condoms plus surgical sterilization (vasectomy at least 1 year prior to enrolment), or
  * Condoms plus surgically sterilised partner (including hysterectomy), or
  * Condoms plus intrauterine device, or
  * Condoms plus partner of non-child bearing potential (including homosexual men) Subjects are required to use condoms to prevent unintended exposure of the partner to the trial drug via seminal fluid.

Alternatively, true abstinence is acceptable when it is in line with the subject's preferred and usual lifestyle. If a subject is usually not sexually active but becomes active, with their partner, they must comply with the contraceptive requirements detailed above.

Exclusion criteria

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 139 mmHg, diastolic blood pressure outside the range of 45 to 89 mmHg, or pulse rate outside the range of 40 to 100 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Clinically significant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/ QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Smoking habit other than incidental. Incidental smoker is defined as a person who will not smoke more than 5 cigarettes per week
* Inability to refrain from smoking in the clinical research unit
* Alcohol abuse (average intake of more than 24 units of alcohol per week (1 unit of alcohol equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits))
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within 96 hours prior to the administration of trial medication and during the trial until the discharge at Day 9
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with trial requirements, or has a condition that would not allow safe participation in the trial

In addition, the following trial-specific exclusion criteria apply:

* A history of chronic kidney disease
* Participation in another absorption, distribution, metabolism, and excretion (ADME) study with a radiation burden of 0.1-1.0 millisievert (mSv) in the period of 1 year prior to screening or 1.1-2.0 mSv in the past 2 years or 2.1-3.0 mSv in the past 3 years etc.
* Exposure to radiation for diagnostic reasons (except dental X-rays and plain X-rays of thorax and bony skeleton (excluding spinal column) in the period of 1 year prior to screening)
* Irregular defecation pattern (less than a mean of one bowel movement every other day)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PRA Health Sciences Onderzoekscentrum Martini, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions: 1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-randomised, open-label, single-dose, single arm, mass balance trial in healthy male subjects.
  The trial had 2 parts. Part 1 was investigating metabolism and pharmacokinetics of (C-14 (radiocarbon labelled)) BI 1265162 after intravenous administration.
  Part 2 was investigating metabolism and pharmacokinetics of (C-14) BI 1265162 after oral administration.
  Part 2 was not conducted due to premature discontinuation of the trial.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- BI 1265162 - Intravenous: Participants received a single intravenous infusion (i.v.) of 50 microgram (μg) of BI 1265162, consisting of 45 μg unlabeled BI 1265162 mixed with 5 μg Carbon 14 labelled BI 1265162 ([14C]BI 1265162) (radocarbon as 10 milliliter (mL) in i.v. solution (5 μg BI 1265162 (C-14)/mL) over 1 hour (h) was administered after an overnight fast of at least 10 h.
  The radioactive dose per infusion was calculated to not exceed 0.018 megabecquerel (MBq).
  Participants received 240 mL of fluid 1 h and 4 h after administration. Participants also received lunch 4 h after administration.
Period: Overall Study
Arm/Group | BI 1265162 - Intravenous
Started | 7
Treated | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set includes all participants who were entered and treated with one dose of trial drug. The treated set will be used for safety analyses.
Arm/Group | BI 1265162 - Intravenous
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.3 (9.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 7
  Female | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Mass Balance Recovery of Total (C-14) BI 1265162-radioactivity in Urine
Description: Mass balance recovery assessed as amount of (C-14) BI 1265162-radioactivity excreted as a percentage of the single intravenous administered dose of BI 1265162 (C-14) over the time interval from 0 to 192 hours.
  The geometric mean and geometric coefficient of variation were calculated by noncompartmental analysis.
Time Frame: On Day -1 or Day 1 pre-dose (blank) sample, on Day 1 prior to start of urine collection voiding of the bladder, 0-4 , 4-8, 8-12, 12-24, 24-48, 48-72, 72-96, 96-120, 120-144, 144-168, and 168-192 hours after administration of BI 1265162 (C-14).
Population: Pharmacokinetic parameter analysis set (PKS): This set includes all participants from the treated set (TS) who provide at least one pharmacokinetic endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of pharmacokinetics or due to pharmacokinetic non-evaluability (as specified in the following subsection 'Pharmacokinetics'). Descriptive analyses of pharmacokinetic parameters will be based on the PKS.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of the administered dose
Arm/Group | BI 1265162 - Intravenous
Number analyzed (Participants) | 7
Percentage of the administered dose | 27.3 (16.1)

2. Primary Outcome: Part 1: Mass Balance Recovery of Total (C-14) BI 1265162-radioactivity in Faeces.
Description: as for outcome 1
Time Frame: On Day -2, Day -1 or Day 1 pre-dose (blank) sample, and on Day 1 0-24, 24-48, 48-72, 72-96, 96-120, 120-144, 144-168, and 168-192 hours after administration of BI 1265162 (C-14).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of the administered dose
Arm/Group | BI 1265162 - Intravenous
Number analyzed (Participants) | 7
Percentage of the administered dose | 65.3 (8.17)

3. Secondary Outcome: Part 1: Area Under the Concentration-time Curve of Total [14C]BI 1265162-equivalent (EQ) in Plasma Over the Time Interval From 0 to 192 Hours (the Last Quantifiable Data Point (AUC0-tz))
Description: Area under the concentration-time curve of total [14C]BI 1265162-EQ in plasma over the time interval from 0 to 192 hours (the last quantifiable data point (AUC0-tz)) was analyzed after the single intravenous dose administration of BI 1265162 (C-14). Plasma concentrations of (C-14) BI 1265162-radioactivity are expressed as [14C]BI 1265162-EQ. The geometric mean and geometric coefficient of variation were calculated by noncompartmental analysis.
Time Frame: At 02:00 hours:minutes pre-dose and at 0:05, 00:30, 00:59 01:05, 01:10, 01:40, 02:00, 03:00, 04:00, 05:00, 07:00, 08:00, 09:00, 11:00, 12:00, 24:00, 48:00, 72:00, 96:00, 120:00, 144:00, 168:00, 192:00 after single dose of BI 1265162 (C-14).
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour times picomole per litre
Arm/Group | BI 1265162 - Intravenous
Number analyzed (Participants) | 7
Hour times picomole per litre | 5290 (27)

4. Secondary Outcome: Part 1: Area Under the Concentration-time Curve of Total BI 1265162 in Plasma Over the Time Interval From 0 to 192 Hours (the Last Quantifiable Data Point (AUC0-tz))
Description: Area under the concentration-time curve of total BI 1265162 in plasma over the time interval from 0 to 192 hours (the last quantifiable data point (AUC0-tz)) was analyzed after the single intravenous dose administration. The geometric mean and geometric coefficient of variation were calculated by noncompartmental analysis.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour times picomole per litre
Arm/Group | BI 1265162 - Intravenous
Number analyzed (Participants) | 7
Hour times picomole per litre | 1890 (12.3)

5. Secondary Outcome: Part 1: Area Under the Concentration-time Curve of Total BI 1265162 Metabolite M582 in Plasma Over the Time Interval From 0 to 192 Hours (the Last Quantifiable Data Point (AUC0-tz))
Description: Area under the concentration-time curve of total BI 1265162 metabolite M582 in plasma over the time interval from 0 to 192 hours (the last quantifiable data point (AUC0-tz)) was analyzed after the single intravenous dose administration. The geometric mean and geometric coefficient of variation were calculated by noncompartmental analysis.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour times picomole per litre
Arm/Group | BI 1265162 - Intravenous
Number analyzed (Participants) | 7
Hour times picomole per litre | 3400 (37.8)

6. Secondary Outcome: Part 1: Maximum Measured Concentration (Cmax) of Total [14C]BI 1265162-equivalent (EQ) in Plasma
Description: Maximum measured concentration (Cmax) of total [14C]BI 1265162-EQ in plasma was analyzed after the single intravenous dose administration. Plasma concentrations of (C-14) BI 1265162-radioactivity are expressed as [14C]BI 1265162-EQ (EQ: equivalent). The geometric mean and geometric coefficient of variation were calculated by noncompartmental analysis.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picomole per litre
Arm/Group | BI 1265162 - Intravenous
Number analyzed (Participants) | 7
Picomole per litre | 2270 (14.7)

7. Secondary Outcome: Part 1: Maximum Measured Concentration (Cmax) of Total BI 1265162 in Plasma
Description: Maximum measured concentration (Cmax) of total BI 1265162 in plasma was analyzed after the single intravenous dose administration. The geometric mean and geometric coefficient of variation were calculated by noncompartmental analysis.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picomole per litre
Arm/Group | BI 1265162 - Intravenous
Number analyzed (Participants) | 7
Picomole per litre | 1880 (15.7)

8. Secondary Outcome: Part 1: Maximum Measured Concentration (Cmax) of Total BI 1265162 Metabolite M582 in Plasma
Description: Maximum measured concentration (Cmax) of total metabolite M582 in plasma was analyzed after single dose administration. The geometric mean and geometric coefficient of variation were calculated by noncompartmental analysis.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picomole per litre
Arm/Group | BI 1265162 - Intravenous
Number analyzed (Participants) | 7
Picomole per litre | 650 (33.9)

9. Secondary Outcome: Part 1: Percentage of Participants With Drug Related Adverse Events (AEs) Including Clinically Relevant Findings From the Physical Examination
Description: Percentage of participants with drug related adverse events (AEs) including clinically relevant findings from the physical examination.
  Percentages are calculated using total number of participants per treatment as the denominator.
Time Frame: From drug administration up to 22 days.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | BI 1265162 - Intravenous
Number analyzed (Participants) | 7
Percentage of participants | 14.3

ADVERSE EVENTS:
Time Frame: From drug administration up to 22 days.
Description: Treated set (TS): The treated set includes all participants who were entered and treated with one dose of trial drug. The treated set will be used for safety analyses.
Arm/Group | BI 1265162 - Intravenous
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 4/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1265162 - Intravenous (N=7)
Toothache (Gastrointestinal disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
The study was interrupted due to COVID-19 crisis on 02-Apr-2020, after completion of Part 1. Further, the sponsor decided to discontinue the development of BI 1265162. Enrolment in Part 2 (oral administration of BI 1265162 (C-14)) did not take place. Decision to terminate trial was taken on 17-Dec-2020.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/76/NCT04267276/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/76/NCT04267276/SAP_001.pdf